CLINICAL TRIAL: NCT04581694
Title: Transcatheter Implantation of Aortic Bioprosthesis Without the Use of Iodinated Contrast in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Fábio Sândoli de Brito Júnior, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FábioSândoli
Record Dates: First submitted 2020-09-25; First posted 2020-10-09 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Stenosis; Valve; Renal Failure; Renal Insufficiency
MeSH Terms: conditions — Constriction, Pathologic; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Twenty-five patients who meet all inclusion criteria and without exclusion criteria will be submitted to TAVI using the "zero contrast" strategy.
  Four imaging methods will be used to evaluate this new strategy: (1) multi-slice computed tomography (TCMS) without contrast, (2) aortoiliac angiography with CO2, (3) nuclear magnetic resonance (MR) of heart without contrast and (4 ) 3D transesophageal echocardiogram (3D TEE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVI without contrast (Experimental)
  Interventions: Diagnostic Test: TAVI without contrast

INTERVENTIONS:
Diagnostic Test: TAVI without contrast — TAVI without contrast

SUMMARY:
Acute renal failure (ARF) after transcatheter aortic valve implantation (TAVI) is a frequent complication, with significant clinical consequences. History of chronic kidney disease and the use of a large amount of iodinated contrast for planning and procedure are among the main risk factors for the development of this complication. The present study aims to: (1) define the role of non-contrast imaging modalities in pre-procedure planning; (2) evaluate the feasibility and safety of a new TAVI technique without using iodinated contrast; (3) to determine the incidence of acute renal failure in patients with aortic stenosis and chronic kidney disease undergoing TAVI, using the new technique without contrast. The study will be divided into two stages. In the pilot phase, 25 consecutive patients with chronic kidney disease (stage ≥ 3a) will have the TAVI planning and procedure performed without the use of iodinated contrast, but with all the steps subjected to verification by the standard technique, to ensure the safety of the patient. The occurrence of the combined primary safety outcome composed of adverse clinical events within 30 days (defined by the VARC-2 criteria) in less than 20% of cases will be used to define the continuity of the study. In the second phase, 50 patients with chronic kidney disease stage ≥ 3b will be submitted to TAVI with the "zero contrast" technique. The primary outcome assessed at this stage of the study will be the incidence of AKI within 7 days after TAVI using the new technique in this high-risk population.

DETAILED DESCRIPTION:
This will be a prospective, single-center, single-arm clinical trial, to be carried out at the Heart Institute of Hospital das Clínicas, Faculty of Medicine, University of São Paulo (InCor - HC - FMUSP). The study will be divided into two phases. The first phase ("pilot") will test the concept, feasibility and safety of using a "zero contrast" strategy to carry out the planning and procedure of TAVI through transfemoral access with the self-expanding bioprosthesis Evolut R / Pro in 25 consecutive patients with CKD. The second phase ("zero contrast") will include 50 patients with CKD who will be submitted to transfemoral TAVI with the Evolut R / Pro bioprosthesis using the "zero contrast" approach, seeking to evaluate the results of the procedure and the incidence of AKI with the new strategy.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with severe aortic valve stenosis (AoS).
* CKD in stage ≥3a (GFR <60mL / min / 1.73m2).
* Signature of the free and informed consent form (ICF).

Exclusion Criteria:

- Any condition considered a contraindication for the implantation of a biological valve prosthesis (for example, the patient has an indication for mechanical valve prosthesis).

• Hypersensitivity or known contraindication to any of the following items that cannot be adequately premedicated: aspirin, clopidogrel or heparin (HIT / HITTS) nitinol (titanium or nickel) the contrast medium (pilot phase)

* Blood dyscrasias: leukopenia (white blood cell count <1000 / mm3), thrombocytopenia (platelet count <50,000 cells / mm3), history of hemorrhagic diathesis, coagulopathy or hypercoagulable states.
* Active infection, including active endocarditis.
* Cardiogenic shock manifested by low cardiac output, dependence on vasopressors or mechanical hemodynamic support.
* Recent stroke (up to 2 months after heart-team evaluation) or transient ischemic attack.
* Gastrointestinal bleeding that prevents platelet anticoagulation or anti-aggregation.
* Refusal to transfuse blood.
* Severe dementia (resulting in the inability to provide informed consent for the study / procedure).
* Life expectancy estimated at less than 12 months.
* Other medical, social or psychological conditions that, in the investigator's opinion, prevent the patient from consenting or adhering adequately to the protocol.
* Pre-existing prosthetic heart valve in the aortic position.
* Presence of stenosis or significant mitral regurgitation.
* Presence of obstructive hypertrophic cardiomyopathy.
* Clinical indication for coronary angiography or percutaneous coronary intervention in the period including the previous 30 days and 30 days after the TAVI procedure. In this case, the use of contrast media for these procedures can be a confusing factor for the analysis of the primary study outcome.
* Contraindication for the transfemoral approach based on evaluation by non-contrast TCMS and by CO2 aortoiliac angiography (anatomical screening).
* High risk of rupture of the ring or significant residual paravalvular leak due to important calcification of the left ventricular outflow tract.
* High risk of coronary occlusion (height of the coronary ostium <10 mm with narrow SOV: <1 mm greater than the size of the bioprosthesis) defined by imaging methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Pilot Phase: Early safety at 30 days - (VARC-2 criteria) | 30 days
  In the pilot phase, we aim to assess the combined primary safety outcome (at 30 days) including all-cause mortality, severe stroke, bleeding with a risk of death, acute renal failure (stages 2 or 3), peri-procedure infarction, major vascular complication and valve-related dysfunction requiring repeated intervention (aortic valvuloplasty, TAVI or surgical valve replacement).
Zero Contrast Phase: incidence of AKI up to a7 days | 7 days
  The incidence of AKI up to 7 days after TAVI will be the primary outcome of the "zero contrast" phase.
  Acute renal failure will be defined according to the VARC-2 criteria and classified into 3 stages:
  * Stage 1: 1.5-1.99-fold increase in serum creatinine compared to baseline OR absolute increase of 0.3 mg / dL OR urine output less than 0.5 mL / kg / h for more than 6 hours, but for less than 12 h;
  * Stage 2: 2.0-2.99-fold increase in serum creatinine compared to baseline OR urine output below 0.5 mL / kg / h for more than 12 hours, but for less than 24 hours;
  * Stage 3: greater than 3-fold increase in serum creatinine compared to baseline OR baseline serum creatinine equal to or greater than 4.0 mg / dL with an acute increase of at least 0.5 mg / dL OR urine output less than 0, 3 mL / kg / h for 24h or more OR anuria for 12h or more. The need for renal replacement therapy, regardless of other criteria, is classified as stage 3 AKI.

SECONDARY OUTCOMES:
Pilot phase: Accuracy in choosing the size of the bioprosthesis. | Procedure - 1 day
  Accuracy in choosing the size of the bioprosthesis based on the non-contrast imaging modalities, compared to the size chosen by another experienced member of the heart-team through the assessment of the contrast-enhanced TCMS, the gold standard method for this purpose. Accuracy is defined as the number of cases with correct choice of the size of the transcatheter prosthesis, divided by the total number of cases treated in the pilot phase.
Pilot phase: Device success (VARC-2 criteria) | Procedure - 1 day
  Success of the device using the "zero contrast" strategy for the TAVI procedure. The device's Absence of death in the procedure AND correct positioning of a single bioprosthesis with the intended performance (mean gradient <20 mmHg and absence of moderate or important aortic insufficiency).
Zero Contrast phase: Device success (VARC-2 criteria) | Procedure - 1 day
  Absence of death in the procedure AND correct positioning of a single bioprosthesis with the intended performance (mean gradient <20 mmHg and absence of moderate or significant aortic insufficiency).
  2. Safety at 30 days: outcome consisting of death from all causes, stroke, bleeding with risk of death, major vascular complication, coronary obstruction, ARF stages 2 or 3, valve-related dysfunction requiring repeated intervention (aortic valvuloplasty) , TAVI or surgical valve replacement)
Zero Contrast phase: Early safety at 30 days - (VARC-2 criteria) | 30 days
  Outcome consisting of death from all causes, stroke, bleeding with risk of death, major vascular complication, coronary obstruction, ARF stages 2 or 3, valve-related dysfunction requiring repeated intervention (aortic valvuloplasty) , TAVI or surgical valve replacement)

CONTACTS AND LOCATIONS:
Overall Officials: Fábio S Brito Jr., PhD, Principal Investigator — Structural Heart Disease - Interventional cardiologist
Locations (1):
- Heart Institute - InCor. University of Sao Paulo Medical School, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided